CLINICAL TRIAL: NCT00259870
Title: A Multi Centre, Double-Blind, Double-Dummy, Placebo-Controlled, Randomised, Adaptive, Dose-Range Study To Evaluate the Safety and Efficacy of SB-773812 Administered Once Daily for 12 Weeks in Adults With Schizophrenia
Brief Title: SB-773812 Administered In Adults With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NAA104606
Record Dates: First submitted 2005-11-30; First posted 2005-12-01 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; PANSS; Acute; Cognition
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SB-773812
Drug: Olanzapine
  Other Names: SB-773812

SUMMARY:
This is a two part study designed to evaluate the safety and efficacy of SB-773812 in the treatment of acute schizophrenia. Subjects with acute schizophrenia will be randomized in an adaptive design study to receive placebo, SB-773812 60mg or olanzapine 15mg for 12 weeks in Part A. An interim analysis will be conducted to assess the efficacy and safety of the SB-773812 60mg dose compared with placebo. Based on these data, up to two further doses of SB-773812 will be added to the randomization for Part B.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for schizophrenia as defined in DSM-IV.
* PANSS total score of at least 70 at Screen and Baseline and a minimum score of 4 (moderate) on at least 2 of the following: conceptual disorganization (P2) hallucinatory behaviour (P3) suspiciousness (P6) or unusual thought content (G9) at the Screen and Baseline visits

Exclusion Criteria:

* Subjects with a history of epilepsy or other seizure disorder, first episode of schizophrenia or other psychotic disorders (e.g. residual type schizophrenia, schizophreniform disorder, schizoaffective disorder, delusional disorder, etc.)
* Bipolar disorder, a history of substance dependence, or a medical or psychiatric disorder that would interfere with the accurate assessment of safety or efficacy are not eligible.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2005-09; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
total score for each SB-773812 dose versus placebo at Week 6. | 12 Weeks

SECONDARY OUTCOMES:
Evaluate safety of SB-773812 versus placebo and compared to olanzapine using PANNS scores -Measure the preliminary pharmacokinetic/pharmacodynamic relationships for SB-773812 -Assessment of movement disorders and cognitive functioning | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (38):
- United States (18):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Cerritos, California
  - GSK Investigational Site, Garden Grove, California
  - GSK Investigational Site, National City, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, North Miami, Florida
  - GSK Investigational Site, Clementon, New Jersey
  - GSK Investigational Site, Kenilworth, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Orangeburg, New York
  - GSK Investigational Site, Butner, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Bellaire, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Falls Church, Virginia
- Belgium (2):
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Montignies-sur-Sambre
- GSK Investigational Site, San José, Costa Rica
- Czechia (3):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Lnáře
  - GSK Investigational Site, Prague
- India (8):
  - GSK Investigational Site, Ahmedabad
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Lucknow
  - GSK Investigational Site, Ludhiana
  - GSK Investigational Site, Mangalore
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Tirupati
- GSK Investigational Site, Lima, Lima Province, Peru
- Russia (5):
  - GSK Investigational Site, Leningraskaya Region
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Smolensk